CLINICAL TRIAL: NCT02092090
Title: A LARGE-SCALE CLUSTER RANDOMIZED TRIAL TO DETERMINE THE EFFECTS OF SODIUM REDUCTION ON STROKE: THE CHINA SALT SUBSTITUTE AND STROKE STUDY (SSaSS)
Brief Title: China Salt Substitute and Stroke Study
Acronym: SSaSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The George Institute (Other)
Collaborators: Peking University (Other); Northwestern University (Other); Imperial College London (Other); China Medical University, China (Other); Changzhi Medical College (Other); Centers for Disease Control and Prevention, China (Other Government); Ningxia Medical University (Other); Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SSaSS; Grant ID 1049417 (Other Grant/Funding Number: Australian National Health and Medical Research Council)
Record Dates: First submitted 2014-03-12; First posted 2014-03-19 (Estimated); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Stroke
Keywords: salt substitute; sodium reduction; stroke; cluster randomized trial; China
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Dietary advice at baseline only
- Dietary sodium reduction (Experimental): Dietary advice and reduced-sodium added-potassium salt substitute
  Interventions: Behavioral: Dietary sodium reduction

INTERVENTIONS:
Behavioral: Dietary sodium reduction — Ongoing dietary advice and a supply of a reduced-sodium added-potassium salt substitute
  Other Names: Reduced-sodium added-potassium salt substitute
  Arms: Dietary sodium reduction

SUMMARY:
The study is a large scale cluster randomised trial to evaluate the effects of sodium reduction based upon the use of salt substitute on the risk of stroke defined as the occurrence of stroke and stroke deaths. The corresponding null hypothesis that will be tested is that sodium reduction will have no effect upon stroke risk. The secondary objectives are to determine effects of sodium reduction on major vascular events and total mortality.

DETAILED DESCRIPTION:
Lowering sodium intake and the use of salt substitute have been proved to lower blood pressure levels. Effects on the risks of vascular outcomes have not been defined in an adequately powered randomised trial. Rural Chinese are known to consume very large quantities of sodium and to suffer from very high rates of hypertension and stroke. This study is a large scale cluster randomised trial done in rural areas of China. The study will define the effects of a salt substitute-based sodium reduction strategy on the primary outcome of stroke. Secondary endpoints will include major cardiovascular events and total mortality. The study will be conducted in 600 rural villages across five Northern Chinese provinces and Tibet. The study will recruit 35 individuals at elevated risk of stroke from each village for a total of 21,000 participants. The participating villages will be randomised into intervention and control group with 1:1 allocation. Recruitment will prioritise individuals with a history of stroke but also include older individuals with high blood pressure. Follow up is scheduled for 5 years. Individuals in intervention villages will receive repeated dietary advice and a supply of low sodium salt substitute while individuals in control villages will receive dietary advice at baseline only. Every 6 months throughout follow-up each individual will be contacted by phone call to inquire about the occurrence of stroke, hospitalisation for any cause and diagnoses of any other serious illnesses. The interview will be structured and done by individuals masked to the randomised assignment of each individual. For all deaths identified and all events that might possibly be non-fatal strokes a home visit will be made. A series of process indicators including urinary sodium, urinary potassium, blood pressure, knowledge about sodium and use of salt substitute will also be measured on a random sample of at least 20 individuals drawn from a random selection of 60 villages at baseline and every year thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Disease history
* Prior stroke and/or
* Aged 60 years or over and with uncontrolled high blood pressure (systolic blood pressure >=140 millimeters of mercury (mmHg) at visit if on blood pressure lowering medication; systolic blood pressure>=160 millimeters of mercury (mmHg) if not on blood pressure lowering medication)
* Ownership of a phone by the participant or a household member

Exclusion Criteria:

* Participant or family member is using a potassium-sparing diuretic
* Participant or family member is using a potassium supplement
* Participant or family member has serious renal impairment
* Participant or family member has other reason for concern about use of salt substitute
* Participant eats most meals outside the home
* Participant is not expected to live longer than 6 months from the date of assessment as estimated by the village doctor
* Another family member living in the same household has already been included in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20996 (Actual)
Dates: Start 2014-07-09 (Actual); Primary Completion 2020-09-04 (Actual); Study Completion 2020-09-04 (Actual)

PRIMARY OUTCOMES:
Stroke | 5 years
  The primary outcome will be stroke defined according to standard criteria on the basis of an acute disturbance of focal neurological function and resulting in death or symptoms lasting more than 24 hours. Imaging, clinical and laboratory data will be collected wherever possible.

SECONDARY OUTCOMES:
Total major vascular events | 5 years
  The composite of stroke, acute coronary syndrome or vascular death
Total mortality | 5 years

OTHER OUTCOMES:
Blood Pressure | 5 years
Urinary sodium excretion | 5 years
Urinary Potassium | 5 years
Knowledge about sodium and salt substitute | 5 years
  Knowledge about sodium and salt substitute will be measured using the following questions at baseline and follow-up:.
  Is a high salt intake good for your health? Does how much salt you eat affect your blood pressure? Does how much salt you eat affect your risk of stroke? What is the daily recommended salt intake for adults? Do you try to reduce the amount of salt you eat? Do you eat pickled vegetables most days? Do you add salt to most meals? Do you add mono-sodium glutamate to most meals? Do you try to eat less of a food if it is very salty? Have you heard about low sodium salt? If yes,does your household use low-sodium salt?

CONTACTS AND LOCATIONS:
Overall Officials: Bruce C Neal, PhD, Principal Investigator — The George Institute for Global Health, Australia; Yangfeng Wu, PhD, Principal Investigator — The George Institute for Global Health at Peking University Health Science Centre; Darwin Labarthe, PhD, Principal Investigator — Northwestern University Feinberg School of Medicine; Paul Elliott, PhD, Principal Investigator — School of Public Health, Imperial College London; Lijing L Yan, PhD, Principal Investigator — The George Institute for Global Health at Peking University Health Science Centre; Nicole Y Li, PhD, Principal Investigator — The George Institute for Global Health, Australia
Locations (5):
- China (5):
  - Hebei Province Centre for Disease Control and Prevention, Shijiazhuang, Hebei
  - China Medical Universtity, Shenyang, Liaoning
  - Ningxia Medical University, Yinchuan, Ningxia
  - Xi'an Jiaotong University, Xi'an, Shaanxi
  - Changzhi Medical Colledge, Changzhi, Shanxi

REFERENCES:
- [Derived] Zhang X, Yin X, Yap ML, Li Q, Huang L, Liu Y, Zhou B, Li Z, Zhao Y, Sun J, Yu Y, Yan LL, Wu Y, Neal B, Tian M. Effect of sodium-reduced potassium-enriched salt substitutes on stomach cancer: the Salt Substitute and Stroke Study (SSaSS). BMC Med. 2025 Apr 23;23(1):236. doi: 10.1186/s12916-025-04068-0. PMID 40264179
- [Derived] Ding X, Zhang X, Huang L, Xiong S, Li Z, Zhao Y, Zhou B, Yin X, Xu B, Wu Y, Neal B, Tian M, Yan LL. Salt Substitution and Recurrent Stroke and Death: A Randomized Clinical Trial. JAMA Cardiol. 2025 Apr 1;10(4):343-350. doi: 10.1001/jamacardio.2024.5417. PMID 39908026
- [Derived] Wang F, Pi Y, Zhao Y, Zhang Y, Zhou B, Li Z, Sun J, Yu Y, Tian M, Yang M, Huang L, Song H, Neal B, Kissock KR. Effect of salt substitution on fracture-a secondary analysis of the Salt Substitute and Stroke Study (SSaSS). BMC Med. 2024 Sep 4;22(1):366. doi: 10.1186/s12916-024-03586-7. PMID 39232779
- [Derived] Yu J, Arnott C, Li Q, Di Tanna GL, Tian M, Huang L, Yin X, Zhang X, Pearson SA, Labarthe DR, Elliott P, Yan LL, Zhou B, Wu Y, Neal B. Secondary Analysis of the Salt Substitute and Stroke Study (SSaSS): Effects of Potassium-Enriched Salt on Cardiac Outcomes. Hypertension. 2024 May;81(5):1031-1040. doi: 10.1161/HYPERTENSIONAHA.123.22410. Epub 2024 Mar 11. PMID 38465623
- [Derived] Haghdoost F, Gnanenthiran SR, Shan S, Kaistha P, Huang L, Tian M, Liu Y, Yin X, Zhang X, Hao Z, Wu Y, Di Tanna GL, Neal B, Rodgers A. The effect of salt substitution on frequency and severity of headache: results from the SSaSS cluster-randomised controlled trial of 20,995 participants. Eur J Clin Nutr. 2024 May;78(5):401-406. doi: 10.1038/s41430-024-01419-7. Epub 2024 Feb 24. PMID 38402353
- [Derived] Yin X, Paige E, Tian M, Li Q, Huang L, Yu J, Rodgers A, Elliott P, Wu Y, Neal B. The Proportion of Dietary Salt Replaced With Potassium-Enriched Salt in the SSaSS: Implications for Scale-Up. Hypertension. 2023 May;80(5):956-965. doi: 10.1161/HYPERTENSIONAHA.122.20115. Epub 2023 Jan 11. PMID 36628969
- [Derived] Neal B, Wu Y, Feng X, Zhang R, Zhang Y, Shi J, Zhang J, Tian M, Huang L, Li Z, Yu Y, Zhao Y, Zhou B, Sun J, Liu Y, Yin X, Hao Z, Yu J, Li KC, Zhang X, Duan P, Wang F, Ma B, Shi W, Di Tanna GL, Stepien S, Shan S, Pearson SA, Li N, Yan LL, Labarthe D, Elliott P. Effect of Salt Substitution on Cardiovascular Events and Death. N Engl J Med. 2021 Sep 16;385(12):1067-1077. doi: 10.1056/NEJMoa2105675. Epub 2021 Aug 29. PMID 34459569
- [Derived] Li KC, Tian M, Neal B, Huang L, Yu J, Liu Y, Yin X, Zhang X, Wu Y, Li N, Elliott P, Yan L, Labarthe D, Hao Z, Shi J, Feng X, Zhang J, Zhang Y, Zhang R, Zhou B, Li Z, Sun J, Zhao Y, Yu Y, Si L, Lung T. Protocol for the economic evaluation of the China Salt Substitute and Stroke Study (SSaSS). BMJ Open. 2021 Jul 20;11(7):e045929. doi: 10.1136/bmjopen-2020-045929. PMID 34285006